CLINICAL TRIAL: NCT05704634
Title: A Phase Ib Study to Evaluate the Safety and Preliminary Efficacy of IL6-receptor Antibody Sarilumab in Combination With antiPD1 Antibody Cemiplimab for Patients With Non-small Cell Lung Cancer.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1194; NCI-2023-00573 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — cemiplimab; sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A : EGFR-mutant cohort (Experimental): Each cohort is planned for 30 Participants with a total of 60 Participants. Participants who are treated in Run-In safety cohort can also be evaluated for efficacy in the molecularly define cohort A or B.
  Interventions: Drug: Cemiplimab; Drug: Kevzara (Sarilumab)
- Cohort B: LKB1-mutant cohort (Experimental): Each cohort is planned for 30 Participants with a total of 60 Participants. Participants who are treated in Run-In safety cohort can also be evaluated for efficacy in the molecularly define cohort A or B.
  Interventions: Drug: Cemiplimab; Drug: Kevzara (Sarilumab)

INTERVENTIONS:
Drug: Cemiplimab — Given by Injection under the skin every 2 weeks
Drug: Kevzara (Sarilumab) — Given by IV (vein) over about 30 minutes every 3 weeks.

SUMMARY:
To learn if the combination of sarilumab (also called Kevzara) and cemiplimab can help to control EGFR- or LKB1/STK11-mutant NSCLC.

DETAILED DESCRIPTION:
Primary Objective:

* To evaluate the safety of sarilumab cemiplimab combination in metastatic lung cancer patients.
* The primary endpoint is DLT for safety Run-In cohort.
* To preliminarily assess efficacy of sarilumab cemiplimab combination in patients with EGFR- or LKB1/STK11-mutant NSCLC respectively.
* The primary efficacy endpoint is objective response rate (ORR) in cohort A and cohort B, evaluated separately.

Secondary Objectives:

--To evaluate the progression-free survival (PFS), disease control rate (DOR), duration of response (DoR), overall survival (OS), and safety and tolerability of this combination in patients with EGFR- or LKB1-mutant NSCLC respectively.

Correlative/Exploratory Objectives:

* Explore the association of baseline genomic profiles (from tumor, germline DNA, and ctDNA) with clinical benefit in patients treated with sarilumab and cemiplimab combination
* Explore the association of immune profiles (tumor immune microenvironment features) with clinical benefit in patients treated with sarilumab and cemiplimab combination
* Explore resistance mechanisms to sarilumab and cemiplimab combination.
* Determine the impact of sarilumab on immunotherapy-related side effects from cemiplimab.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Histologically or cytologically confirmed non-squamous, non-small cell lung cancer
4. Locally advanced or metastatic disease.
5. Patients must have one of the following:

   Cohort A:
   * NSCLC which harbours EGFR Exon 19 deletion.
   * NSCLC which harbours EGFR L858R mutation.
   * NSCLC with activating EGFR exon20 insertion or exon 18/21 atypical mutations EGFR deletion/mutation must be documented by a Clinical Laboratory Improvement Amendments (CLIA) certified test (either from tissue or ctDNA from blood is allowed)

   The documentation of EGFR mutation status can be obtained any time since the initial diagnosis of non-small cell lung cancer.

   For cohort A, the patient must have received an EGFR TKI treatment, if approval targeted therapy exists.

   For patients whose tumor harboring EGFR Exon19 deletion or L858R mutation, prior osimertinib treatment is required, unless contraindicated for medical reasons.

   Cohort B:

   • NSCLC which harbours LKB1 mutation. LKB1 mutation must be documented by a Clinical Laboratory Improvement Amendments (CLIA) certified test (either from tissue or ctDNA from blood is allowed) The documentation of LKB1 mutation status can be obtained any time since the initial diagnosis of non-small cell lung cancer.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Appendix A)
7. At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline at equal or greater than 10mm in the longest dimension by RECIST 1.1.
8. Prior treatment with cytotoxic chemotherapy or immunotherapy is allowed for both cohorts. Up to 3 lines of prior therapy is allowed.
9. Patients must have adequate hematologic, coagulation, hepatic, and renal function. All laboratory tests must be obtained less than 4 weeks from study entry. This includes:

   * ANC >/= 2,000/mm3 and white blood cells >/= 3,000/mm3
   * platelet count >/=150,000/mm3
   * HgB ≥ 8.5 g/dL
   * Creatinine ≤ 30 mL/minute (using Cockroft-Gault formula).
   * Total Serum Bilirubin ≤ ULN (unless with documented Gilbert Syndrome diagnosed by genetic testing)
   * SGOT, SGPT ≤ 1.5 X ULN
   * Cholestrol ≤ 350 mg/dL, 9.1 mmol/L, and triglyceride ≤ 500 mg/dL, 5.6 mmol/.
10. Females of childbearing potential must not be breast feeding and must have a negative serum or urine pregnancy test within 7 days of starting of treatment. The patient must agree to use adequate contraception for a minimum of two weeks prior to receiving study medication until 3 months after discontinuation of the study medication. Acceptable methods of contraception include total and true sexual abstinence, hormonal contraceptives that are not prone to drug-drug interactions (IUS Levonorgestrel Intra Uterine System (Mirena), Medroxyprogesterone injections (Depo-Provera)), copper-banded intra-uterine devices, and vasectomized partner. All hormonal methods of contraception should be used in combination with the use of a condom by their sexual male partner. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause). Women will be considered post-menopausal if they have been amenorrheic for the past 12 months without an alternative medical cause. The following age-specific requirements must also apply: Women < 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of exogenous hormonal treatments. The levels of Luteinizing Hormone (LH) and Follicle-Stimulating Hormone (FSH) must also be in the post-menopausal range (as per the institution). Women ≥ 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of all exogenous hormonal treatments, or have had radiation-induced oophorectomy with the last menses > 1 year ago, or have had chemotherapy-induced menopause with >1 year interval since last menses, or have had surgical sterilization by either bilateral oophorectomy or hysterectomy.
11. Non-sterilized males who are sexually active with a female partner of childbearing potential must use adequate contraception for the duration of the study and 3 months after the last dose of study medication. Adequate contraception methods include: birth control pills (e.g. combined oral contraceptive pill), barrier protection (e.g. condom plus spermicide, cervical/vault cap or intrauterine device), and abstinence. Patients should not father a child for 6 months after completion of the study medication. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing the study medication. If male patients wish to father children they should be advised to arrange for freezing of sperm samples prior to the start of the study medication.
12. Patients who meet eligibility criteria to either Cohort A or B will be allowed to enroll to the run-in cohort.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Spinal cord compression or brain metastases unless asymptomatic or stable for at least 2 weeks prior to start of study treatment.
2. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 (with the exception of alopecia grade 2) at the time of starting study treatment.
3. Any evidence of severe or uncontrolled systemic diseases. Screening for chronic conditions is not required.
4. Woman of childbearing potential (WOCBP) not protected by highly-effective contraceptive method(s) of birth control, and/or who are unwilling or unable to be tested for pregnancy.
5. Pregnant or breastfeeding woman
6. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirement.
7. Active or severe autoimmune disorders, including rheumatoid arthritis
8. Exclusion related to Tuberculosis (TB):

   * Active TB or a history of incompletely treated TB regardless of screening Quantiferon result
   * Quantiferon positive patients (no active disease) are excluded from the study unless the following conditions are met:
   * Patients with a history of prior documented completed chemoprophylaxis for latent tuberculosis infection (eg, acceptable treatments include 9 months of isoniazid 300 mg oral daily or equivalent proven regimen per local guidelines) or treatment of active tuberculosis infection (TBI) who has obtained consultation with a specialist to rule out active TBI or the need to receive further treatment.
   * Patients with no prior history of chemoprophylaxis for latent TBI or treatment for active TBI but have obtained consultation with a specialist to initiate an appropriate regimen of chemoprophylaxis, based on local epidemiology and applicable guidelines and have demonstrated compliance and tolerated treatment for 1 month.

   Consultations with and prior approval from IND sponsor are required in either of the aforementioned scenarios.
   * Clinically significant abnormality consistent with prior/active TB infection based upon chest radiograph with at least posterior-anterior view (See Section 10.8.1). Additional lateral view is recommended but not required.
   * Suspected extra-pulmonary TB infection regardless of screening Quantiferon result.
   * Patients at high risk of contracting TB, such as close contact with individuals with active or latent TB.
   * Patient who received Bacille Calmette Guerin -vaccination within 12 months prior to screening.
9. Patients with a history of invasive opportunistic infections, including but not limited to histoplasmosis, listeriosis, coccidioidomycosis, candidiasis, pneumocystis jirovecii, aspergillosis despite resolution or John Cunningham virus (progressive multifocal leukoencephalopathy).
10. Patients with fever (>38°C) associated with infection, or chronic, persistent, or recurring infection(s) requiring active treatment with antibiotics, antivirals, or antifungals within 4 weeks prior to the screening visit or other frequent recurrent infections deemed unacceptable as per Investigator judgment.
11. Patients with uncontrolled diabetes mellitus, defined as glycosylated hemoglobin (HbA1c) greater than 9% at the screening visit.
12. Patients with non-healed or healing skin ulcers.
13. Patients who received any live, attenuated vaccine within 3 months prior to the baseline visit, such as varicella-zoster, oral polio or rubella vaccines.
14. Patients who are positive for hepatitis B surface antigen (HBsAg) or are positive for total hepatitis B core antibody (HBcAb) with negative hepatitis B surface antibody (HBsAb) or are positive for both HBcAb and HBsAb with presence of HBV DNA at screening. E 25. Patients who are positive for hepatitis C antibody (HCV Ab).
15. Patients who are positive for human immunodeficiency virus (HIV) antibody test at screening or who previously had a positive HIV antibody test, or who are suspected to be positive for HIV.
16. Patients with a history of recurrent herpes zoster or active herpes zoster.
17. Patients with a history of prior articular or prosthetic joint infection.
18. Prior or current history of malignancy, including lymphoproliferative diseases, other than adequately treated carcinoma in-situ of the cervix, non-metastatic squamous cell or basal cell carcinoma of the skin, within 5 years prior to the baseline visit.
19. Prior or current history of other significant concomitant illness(es) that, according to Investigator's judgment, would adversely affect the patient's participation in the study. These include, but are not limited to, cardiovascular (including Stage III or IV cardiac failure according to the New York Heart Association classification), renal, neurological (including demyelinating disease), active infectious diseases, endocrinological, gastrointestinal, hepato-biliary, metabolic, pulmonary, non-malignant lymphoproliferative disease or other lymphatic disease(s).
20. Patients who have had surgery within 4 weeks prior to the screening visit or with planned surgery during the course of the study.
21. Patients with a history of a systemic hypersensitivity reaction, other than localized injection site reaction, to any biologic drug and known hypersensitivity to any constituent of the sarilumab product.
22. Patients with a history of inflammatory bowel disease or severe diverticulitis or previous gastrointestinal perforation.
23. Cognitively impaired adults.
24. Uncontrolled or significant heart disease, such as long QTc interval greater than 480ms on baseline EKG, NYHA III/IV heart failure or uncontrolled arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiuning Le, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org